CLINICAL TRIAL: NCT02625844
Title: Croatian Time and Motion Survey for Anaemia Management With Erythropoietin Stimulating Agents in Haemodialysis Units
Brief Title: Health Care Personnel Time for Anemia Management With Erythropoiesis Stimulating Agents in Hemodialysis Centers in Croatia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25720
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Renal Anemia of Chronic Kidney Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Monopegylated Epoetin Beta: Health care personnel performing anemia management tasks for patients using monopegylated epoetin beta.
  Interventions: Other: No intervention
- Other Erythropoiesis Stimulating Agents (ESAs): Health care personnel performing anemia management tasks for patients using other ESAs.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study.

SUMMARY:
This study is to document the time spent by health care personnel on anemia-related tasks, including preparation, distribution and administration of monopegylated epoetin beta (Mircera) or other erythropoiesis-stimulating agents (ESAs) in patients with end stage renal disease in hemodialysis centers in Croatia. The total average time will be determined for the same number of patients on monopegylated epoetin beta and patients on other ESAs. In addition, qualitative information will be obtained on changes in practice patterns that may have occurred with the introduction of monopegylated epoetin beta.

ELIGIBILITY:
Inclusion Criteria:

- Treatment of symptomatic anemia associated with chronic kidney disease (CKD) in adult patients

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health care personnel providing care for patients with renal anemia on monopegylated epoetin beta or other erythropoiesis stimulating agents (ESAs)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Croatia (4):
  - Bjelovar
  - Split
  - Zadar
  - Zagreb

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient disposition information was unavailable. Therefore, all participants are represented in one arm.
Groups:
- Erythropoiesis Stimulating Agents (ESAs): Healthcare personnel performing anemia care for patients.
Period: Overall Study
Arm/Group | Erythropoiesis Stimulating Agents (ESAs)
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erythropoiesis Stimulating Agents (ESAs)
Number analyzed (Participants) | 110
Age, Customized [Number; unit: participants]
  >/= 18 years | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Gender data were not collected for study participants.
  Male | NA — Gender data were not collected for study participants.

OUTCOME MEASURES:

1. Primary Outcome: Average Observed Health Care Personnel Time for Anemia Management With Erythropoiesis Stimulating Agents (ESAs)
Description: Health care personnel time (hours/year) includes preparation, distribution and administration of Erythropoiesis Stimulating Agents (ESAs)
Time Frame: Up to 3 months
Measure: Number; unit: hours/year
Arm/Group | Erythropoiesis Stimulating Agents (ESAs)
Number analyzed (Participants) | 110
hours/year
  Monopegylated Site 1 | 38
  Monopegylated Site 2 | 15
  Monopegylated Site 3 | 17
  Monopegylated Site 4 | 5
  Other ESAs Site 1 | 143
  Other ESAs Site 2 | 39
  Other ESAs Site 3 | 48
  Other ESAs Site 4 | 22

ADVERSE EVENTS:
Description: Adverse events were not collected for this study.
Arm/Group | Erythropoiesis Stimulating Agents (ESAs)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.